CLINICAL TRIAL: NCT02800330
Title: The Effects of the Proton Pump Inhibitor Esomeprazole on the Bioavailability of Regorafenib in Patients With Metastatic Colorectal Cancer (mCRC) or Gastrointestinal Stromal Tumour (GIST)
Brief Title: The Effects of the Proton Pump Inhibitor Esomeprazole on the Bioavailability of Regorafenib
Acronym: REGORA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Prof. R.H.J. Mathijssen, MD, PhD, Prof, MD, PhD, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EMC16-165
Record Dates: First submitted 2016-05-25; First posted 2016-06-15 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Neoplasms; Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Colorectal Neoplasms; Gastrointestinal Stromal Tumors | interventions — Esomeprazole; Lead; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (e.g. sequence phase A-B-C) (Other): In this arm patients will use regorafenib alone in the first cycle (treatment A), then regorafenib with esomeprazole concomitantly in the second cycle (treatment B) and at last they will use regorafenib with esomeprazole 3 hours before (treatment C)
  Interventions: Drug: Esomeprazole 40mg concomitantly; Drug: Esomeprazole 40mg before; Drug: Regorafenib 160mg or 120mg
- Arm B (e.q. sequence phase C-B-A) (Other): In this arm patients will use regorafenib with esomeprazole 3 hours before (treatment C), then regorafenib with esomeprazole concomitantly in the second cycle (treatment B) and at last they will use regorafenib alone (treatment A),
  Interventions: Drug: Esomeprazole 40mg concomitantly; Drug: Esomeprazole 40mg before; Drug: Regorafenib 160mg or 120mg

INTERVENTIONS:
Drug: Esomeprazole 40mg concomitantly — During phase B the patients will use esomeprazole 40mg concomitantly with regorafenib for 5 days.
  Other Names: phase B
Drug: Esomeprazole 40mg before — During phase C the patients will use esomeprazole 40mg 3 hours before regorafenib for 5 days.
  Other Names: phase C
Drug: Regorafenib 160mg or 120mg — Patients will use regorafenib 160mg or 120mg during all phases (A, B, C)

SUMMARY:
Regorafenib is a novel oral multi-kinase inhibitor which targets angiogenic, stromal and oncogenic receptor tyrosine kinases. It is currently registered for GIST and mCRC. When regorafenib is co-administered with an acid suppressive agent, the intra-gastric pH increases, and as a result the equilibrium of ionized/non-ionized regorafenib may shift to the less soluble non-ionized form which reduces regorafenib bioavailability and exposure. Since proton pump inhibitors (PPIs) are often used during regorafenib therapy, this drug-drug interaction (DDI) confronts pharmacists and oncologists with challenges in clinical practice. In this study the investigators will therefore evaluate the impact of PPI-induced intra-gastric pH elevation on regorafenib pharmacokinetics in patients with GIST and mCRC.

DETAILED DESCRIPTION:
Patients will start with regorafenib in a loading phase of 21 days and will be admitted for 24 hours to the hospital for pharmacokinetic blood sampling on day 21, 49 and 77 (± 1-2 days). Patients will be randomized into 2 sequence groups (respectively sequences phase A-B-C or phase C-B-A). The patient will use regorafenib alone (phase A) or with esomeprazole for five days (phases B and C). To (completely) rule out a pH-dependent DDI between regorafenib and esomeprazole, during phase B of the study regorafenib is given concomitantly for five days, while during phase C regorafenib is given 3 hours after esomeprazole intake for five days (when the intragastric pH is maximally elevated by esomeprazole).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histological or cytological confirmed diagnosis of mCRC or GIST and prior treatment specific:

   1. mCRC-patients who have been previously treated with, or are not considered candidates for, available therapies according to common practice.
   2. Irresectable or metastatic GIST who progressed on or are intolerant to prior treatment with imatinib and sunitinib.
3. ECOG Performance Status ≤ 1
4. Able and willing to sign the Informed Consent Form
5. No concurrent (over the counter) use of other acid reducing drugs (PPIs, H2As and/or antacids), other than esomeprazole 40mg once daily during the study.
6. No concurrent medication or supplements which can interact with esomeprazole or regorafenib during the study period.
7. Abstain from grapefruit, grapefruit juice, herbal dietary supplements, and herbal tea during the study period.
8. Adequate baseline patient characteristics (complete blood count, and serum biochemistry which involves sodium, potassium, creatinin, calculation of creatinin clearance (MDRD), AST, ALT, gamma glutamyl transpeptidase, lipase, lactate dehydrogenase, ALP, total bilirubin, albumin, glucose, INR, thyroid function tests, and PTT or APTT within two weeks prior to the study).

Exclusion Criteria:

1. Pregnant or lactating patients.
2. Patients with known impaired drug absorption (e.g. gastrectomy and achlorhydria).
3. Known serious illness or medical unstable conditions that could interfere with this study; requiring treatment (e.g. infection, bleedings, uncontrolled hypertension despite optimal medical management, HIV, hepatitis, organ transplants, kidney, cardiac and respiratory diseases).
4. Non-healing wound, non-healing ulcer, or non-healing bone fracture
5. Major surgical procedure or significant traumatic injury within 28 days before start of study medication.
6. Patients with evidence or history of any bleeding diathesis, irrespective of severity
7. Any hemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of study medication.
8. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 month before the start of study medication (except for adequately treated catheter-related venous thrombosis occurring more than one month before the start of study medication)
9. Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months)
10. Myocardial infarction less than 6 months before start of study drug.
11. Uncontrolled cardiac arrhythmias
12. Symptomatic CNS metastases or history of psychiatric disorder that would prohibit the understanding and giving of informed consent.
13. Interstitial lung disease with ongoing signs and symptoms at the time of informed consent
14. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation.
15. Known history of HIV infection, active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy.
16. Patients on strong CYP3A4 inhibitors or inducers are not eligible for the study (see appendix B).
17. The use of BCRP or P-glycoprotein substrates which leads to a clinically relevant drug-drug interaction concerning the pharmacokinetics of regorafenib.
18. Unwillingness to abstain from grapefruit (juice), (herbal) dietary supplements, herbals, over-the-counter medication (except for paracetamol and ibuprofen) and other drugs known to seriously interact with esomeprazole and regorafenib during the study period.
19. Unwillingness to abstain from acid beverages such as orange juice and other acidic beverages (e.g. Coca-Cola, 7-UP etc.) in the morning (between 06.00-14.00u AM) during regorafenib treatment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-05; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
As primary endpoint, AUC of regorafenib alone and AUC of regorafenib with esomeprazole (concomitantly and 3 hours before regorafenib intake, respectively) will be related. | T=0, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 6h, 8h, 12h, 24h at day 21, day 49 and day 77
  The AUC of regorafenib will be determined by multiple blood samples at T=0, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 6h, 8h, 12h, 24h at day 21, day 49 and day 77

SECONDARY OUTCOMES:
The Cmax of regorafenib alone and regorafenib with esomeprazole (concomitantly and 3 hours before regorafenib intake respectively) will be related | T=0, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 6h, 8h, 12h, 24h at day 21, day 49 and day 77
  The Cmax of regorafenib will be determined by multiple blood samples at T=0, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 6h, 8h, 12h, 24h at day 21, day 49 and day 77
Number of participants with treatment related adverse events as assessed by CTCAE v4.0 in absence and presence of esomeprazole | Through study completion, approximately 0.5 year
The Tmax of regorafenib alone and regorafenib with esomeprazole (concomitantly and 3 hours before regorafenib intake respectively) will be related | T=0, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 6h, 8h, 12h, 24h at day 21, day 49 and day 77
  The Tmax of regorafenib will be determined by multiple blood samples at T=0, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 6h, 8h, 12h, 24h at day 21, day 49 and day 77
The clearance of regorafenib alone and regorafenib with esomeprazole (concomitantly and 3 hours before regorafenib intake respectively) will be related | T=0, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 6h, 8h, 12h, 24h at day 21, day 49 and day 77
  The clearance of regorafenib will be determined by multiple blood samples at T=0, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 6h, 8h, 12h, 24h at day 21, day 49 and day 77

CONTACTS AND LOCATIONS:
Overall Officials: R.H.J. Mathijssen, MD, PhD, Principal Investigator — EMC
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided